CLINICAL TRIAL: NCT02128061
Title: Sub-cutaneous Rituximab-miniCHOP Versus Sub-cutaneous Rituximab-miniCHOP + Lenalidomide (R2-miniCHOP) in Diffuse Large B Cell Lymphoma for Patients of 80 Years Old or More. A Multicentric Phase III Study of the LYSA Association
Brief Title: Efficacy of Lenalidomide in Combination With Subcutaneous Rituximab + miniCHOP in DLBCL Patients of 80 y/o or+
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Collaborators: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SENIOR
Record Dates: First submitted 2014-04-23; First posted 2014-05-01 (Estimated); Last update posted 2021-04-13 (Actual); Status verified 2020-03

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Lenalidomide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- R-miniCHOP (Active Comparator): All patients will be treated with R-miniCHOP at a three-weeks interval for 6 cycles CYCLOPHOSPHAMIDE IV: 400 mg/m² Day 1 (D1) DOXORUBICINE IV : 25 mg/m² D1 VINCRISTINE IV : 1 mg Total Dose (TD) D1 PREDNISONE PO : 40 mg/m² D1 to D5 RITUXIMAB SC* : 1400 mg TD D1
  *The first cycle of rituximab is delivered by IV at the dose of 375 mg/m2
  Interventions: Drug: Rituximab
- R2-miniCHOP (Experimental): All patients will be treated with R2-miniCHOP at a three-weeks interval for 6 cycles CYCLOPHOSPHAMIDE IV: 400 mg/m² D1 - DOXORUBICINE IV : 25 mg/m² D1 - VINCRISTINE IV : 1 mg TD D1 - PREDNISONE PO : 40 mg/m² D1 to D5 - RITUXIMAB SC* : 1400 mg TD D1 LENALIDOMIDE PO** :10 mg TD D1 to D14
  *The first cycle of rituximab is delivered by IV at the dose of 375 mg/m2
  Interventions: Drug: Lenalidomide; Drug: Rituximab

INTERVENTIONS:
Drug: Lenalidomide
  Other Names: Revlimid
  Arms: R2-miniCHOP
Drug: Rituximab
  Other Names: Mabthera

SUMMARY:
The purpose of this study is to compare the efficacy of R2-miniCHOP (Sub-cutaneous Rituximab-miniCHOP + lenalidomide) and R-miniCHOP (Sub-cutaneous Rituximab-miniCHOP) in patients aged 80 years old or more with not previously treated cluster of differentiation antigen 20 positive (CD20+) diffuse large B-cell lymphoma as measured by the overall survival (OS).The SENIOR trial will evaluate the tolerance and efficacy of the combination of the R2-miniCHOP regimen and compare this experimental arm to the standard R-miniCHOP regimen.The statistical plan is based on the hypothesis of an increase by 15% of the 2y-OS in favor of the experimental arm, as compared to the reference arm (R-miniCHOP).

DETAILED DESCRIPTION:
The purpose of this study is to compare the efficacy of R2-miniCHOP (Sub-cutaneous Rituximab-miniCHOP + lenalidomide) and R-miniCHOP (Sub-cutaneous Rituximab-miniCHOP) in patients aged 80 years old or more with not previously treated cluster of differentiation antigen 20 positive (CD20+) diffuse large B-cell lymphoma as measured by the overall survival (OS).

Primary endpoint of the study is to compare the efficacy of R2-miniCHOP (Sub-cutaneous Rituximab-miniCHOP + lenalidomide) and R-miniCHOP ((Sub-cutaneous Rituximab-miniCHOP) in patients of 80 years old or more with not previously treated CD20+ diffuse large B-cell lymphoma as measured by the overall survival (OS).

Secondary endpoints are:

* To evaluate the efficacy and the safety of R2-miniCHOP as measured by the PFS (Progression Free Survival), EFS (Event Free Survival), the DoR (duration of response), the DFS (disease free survival), response rate at the end of the treatment, the additional toxicities
* To evaluate the simplified scale prognostic impact (IADL, MNA, G8, CIRS-G)
* To assess the quality of life before and after treatment This study is a multicentric, phase III, open-label, randomized (1:1) trial evaluating the efficacy of R2-miniCHOP in patients aged of 80 years or more with non-previously treated CD20+ diffuse large B-cell lymphoma (age-adjusted IPI= 0 to 3), Ann Arbor stage II to IV with a performance status ECOG from 0 to 2.

This study includes a run in phase to assess feasibility, safety and tolerance of subcutaneous rituximab injections and oral lenalidomide (10 mg D1-D14) in combination with dose-reduced intensity CHOP regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically proven CD20+ diffuse large B-cell lymphoma (DLBCL) (WHO classification 2008) including all clinical subtypes (primary mediastinal, intravascular, etc…), with all age-adjusted International Prognostic Index (aaIPI).

May also be included: De Novo transformed DLBCL from low grade lymphoma (Follicular, other...) and DLBCL associated with some small cell Infiltration in bone marrow or lymph node; or CD20+ B-cell lymphoma, with intermediate features between DLBCL and Burkitt or with intermediate features between DLBCL and classical Hodgkin lymphoma; or CD20+ Follicular lymphoma grade 3B (according to WHO classification); or CD20+ Aggressive B-cell lymphoma unclassifiable.

* With a Cluster of Differentiation antigen 10 (CD10) immunostaining performed by the participating center pathologist
* Aged ≥ 80 years old
* Ann Arbor stage II, III or IV
* Patient previously untreated for DLBCL Lymphoma
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* With a minimum life expectancy of 3 months
* Negative HIV, HBV and HCV serologies test within 4 weeks before inclusion (except after hepatitis B vaccination or for patients who are HBs Ag negative, anti-HBs positive and/or anti-HBc positive but viral DNA negative)
* Patient able to give his consent and having signed a written Informed consent
* Patient affiliated to social security system, if applicable
* Male patients must practice complete abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions, and for 3 months following study drug discontinuation, even if they have undergone a successful vasectomy.
* All patients must agree to fulfill the global Lenalidomide Pregnancy Prevention Risk Management Plan as applicable according to the randomization arm (randomization arm)

Exclusion Criteria:

* Any other histological type of lymphoma, Burkitt included
* Any history of treated or non-treated small-B cell lymphoma
* Central nervous system or meningeal involvement by lymphoma
* Contra-indication to any drug contained in the chemotherapy regimens ; for anthracycline use, ejection fraction should be > 50%
* Any serious active disease (according to the investigator's decision)
* History of deep venous thrombosis or arterial thromboembolism events within the past 12 months before inclusion
* Poor renal function (creatinine clearance < 40 ml/min, according to Modification of Diet in Renal Disease (MDRD) formula)
* Poor hepatic function (total bilirubin level >30mmol/l, transaminases >2.5 maximum normal level) unless these abnormalities are related to the lymphoma
* Poor bone marrow reserve as defined by neutrophils <1.5 G/l or platelets <100 G/l, unless related to bone marrow infiltration
* Any history of cancer during the last 5 years with the exception of non-melanoma skin tumors or stage 0 (in situ) cervical carcinoma Patients previously diagnosed with prostate cancer are eligible if (1) their disease was T1-T2a, N0, M0, with a Gleason score ≤7, and a prostate specific antigen (PSA) ≤10 ng/mL prior to initial therapy, (2) they had definitive curative therapy (i.e., prostatectomy or radiotherapy) 2 years before Day 1 of Cycle 1, and (3) at a minimum 2 years following therapy they had no clinical evidence of prostate cancer, and their PSA was undetectable if they underwent prostatectomy or <1 ng/mL if they did not undergo prostatectomy
* Treatment with any investigational drug within 30 days before planned first cycle of chemotherapy and during the study
* Prior treatment with anti-CD20 monoclonal antibody or alemtuzumab within 3 months prior to start of therapy
* Prior use of lenalidomide
* Prior ≥ Grade 3 allergic reaction/hypersensitivity to thalidomide
* Prior ≥ Grade 3 rash or any desquamating (blistering) rash while taking thalidomide
* Subjects with ≥ Grade 2 neuropathy
* Adult patient under tutelage
* Female of childbearing potential are excluded. (Note: Females are defined as not of childbearing potential if there is documentation of "natural menopause for at least 24 consecutive months, a hysterectomy or bilateral oophorectomy")

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 250 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
The overall survival (OS) | OS rates at 2 years
  OS will be measured from the date of randomization to the date of death from any cause. Alive patients will be censored at their last contact.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | PFS rates at 2 years
  PFS is defined as the time from randomization into the study to the first observation of documented disease progression/relapse or death due to any cause. If a subject has not progressed or died, PFS will be censored at the time of last visit with adequate assessment.
Event-Free Survival (EFS) | EFS rates at 2 years
  EFS will be measured from the date of randomization to the date of first documented disease progression/relapse (Cheson 1999), initiation of new anti-lymphoma therapy or death from any cause. Patients without documented event at the time of analysis will be censored at their visit with adequate assessment.
Duration of Response (DoR) | DoR rates at 2 years
  DoR will be measured from the time of attainment of Complete Response/unconfirmed Complete Response (CR/CRu) or Partial Response (PR) to the date of first documented disease progression/relapse or death from any cause. Patients alive and free of progression will be censored at their last visit with adequate assessment.
Disease-Free Survival (DFS) | DFS rates at 2 years
  DFS will be measured from the date of attainment of a complete or unconfirmed complete response (at the end of treatment or at permanent treatment discontinuation evaluation) to the date of first observation of documented disease progression or death due to any cause. Complete Response/unconfirmed Complete Response (CR/CRu) patients who have not progressed or died will be censored at the time of last visit with adequate assessment.
OS according to GCB/non-GCB phenotype | OS according to GCB/non-GCB phenotype rates at 2 years
  OS will be described for the R2-miniCHOP group according to Hans algorithm (GCB/non-GCB phenotype).
Response Rate at the end of treatment | 22 weeks (28 days after the end of the 6, three-weeks interval, cycles of treatment) or within 28 days following permanent treatment discontinuation
  Disease response evaluation at end of treatment (after 6 cycles) will be used to determine the Response Rate. Response will be assessed at end of treatment (after end of the 6th cycle of treatment or at permanent treatment discontinuation).
  Assessment of response will be based on the International Workshop to Standardize Response criteria for non-Hodgkin's lymphoma (NHL) (Criteria for evaluation of response in NHL (Cheson, 1999)).
Simplified Geriatric Scales | At baseline
  Four geriatric tools will be performed before any chemotherapy administration (Instrumental Activities of Daily Living (IADL), Mini Nutritional Assessment (MNA), G8, and Cumulative Illness Rating Scale for Geriatrics (CIRS-G) scales). Each scale will be analyzed in order to have a picture of the population at baseline. Thereafter, the prognosis impact in OS and PFS of each scale will be evaluated using univariate (Kaplan Meier) and multivariate analyses (Cox model). Safety analyses will also be performed according to each scale in order to evaluate the toxicity predictive power of these scales.
Health related Quality of Life (HRQOL) | At randomization and 22 weeks after Day 1 of Cycle 1 of R-miniCHOP or R2-miniCHOP (28 days after the end of the 6, three-weeks interval, cycles of treatment)
  HRQOL will be assessed by the Quality of Life Questionnaire-C30 and Elderly14 (QLQ-C30 and the QLQ-ELD14) at randomization and at end of treatment. The improvement or not of the QoL will therefore be assessed.
  The QLQ-ELD14 was developed to supplement the QLQ-C30 for measuring HRQoL in patients aged >70 years in oncology studies.

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Jardin, MD,Professor, Principal Investigator — The Lymphoma Study Association - LYSA
Locations (97):
- Belgium (14):
  - ZNA Stuivenberg, Antwerp
  - A. Z. Sint-Jan, Bruges
  - Institut Jules Bordet, Brussels
  - Université Catholique de Louvain Saint Luc, Brussels
  - Hôpital Erasme, Brussels
  - Grand Hôpital de Charleroi, Charleroi
  - Universitair Ziekenhuis Gent, Ghent
  - AZ Groeninge, Kortrijk
  - CHR Citadelle, Liège
  - CHU de Liège, Liège
  - Hôpital Sainte Elisabeth, Namur
  - Clinique Saint Pierre, Ottignies
  - CHR Peltzer La Tourelle, Verviers
  - CHRU Mont Godinne, Yvoir
- France (83):
  - CH d'Abbeville, Abbeville
  - CH du Pays d'Aix, Aix-en-Provence
  - CHU d'Amiens, Amiens
  - CHU d'Angers, Angers
  - CH Victor Dupouy, Argenteuil
  - CH d'Arras, Arras
  - CH d Avignon - Hopital Henri Duffaut, Avignon
  - CH Côte Basque, Bayonne
  - CHU Jean Minjoz, Besançon
  - CH de Blois, Blois
  - Institut Bergonié, Bordeaux
  - Polyclinique Bordeaux Nord, Bordeaux
  - CH de Boulogne-sur-Mer, Boulogne-sur-Mer
  - CH de Bourg en Bresse, Bourg-en-Bresse
  - CHU Morvan, Brest
  - CH de Brive, Brivé
  - IHBN, Caen
  - CH de Cannes, Cannes
  - Clinique Du Parc, Castelnau-le-Lez
  - Médipôle de Savoie, Challes-les-Eaux
  - CHU de Châlon sur Sâone, Chalon-sur-Sâone
  - CH Métropole Savoie, Chambéry
  - Hôpital d'Instruction des Armées Percy, Clamart
  - CHU Estaing, Clermont-Ferrand
  - Pôle Santé République, Clermont-Ferrand
  - CH Sud Francilien de Corbeil, Corbeil-Essonnes
  - APHP - Hopital Henri Mondor, Créteil
  - CHU de Dijon - Hôpital le Bocage, Dijon
  - CH de Dunkerque, Dunkirk
  - CH Eure Seine, Évreux
  - CHU de Grenoble, Grenoble
  - Institut Daniel Hollard, Grenoble
  - CH Départemental de Vendée, La Roche-sur-Yon
  - Hôpital St Louis, La Rochelle
  - CH de Versailles - Hopital André Mignot, Le Chesnay
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CH du Mans, Le Mans
  - Clinique Victor Hugo, Le Mans
  - CHRU Lille - Hôpital Claude Huriez, Lille
  - Hôpital Saint Vincent de Paul, Lille
  - CHU de Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmette, Marseille
  - Hôpital de la conception, Marseille
  - CH des Chanaux, Mâcon
  - CH de Meaux, Meaux
  - Hôpital de Mercy, Metz
  - Centre Hospitalier Annecy Genevois, Metz-Tessy
  - CHU de Montpellier, Montpellier
  - CHU de Mulhouse, Mulhouse
  - CHU de Nantes, Nantes
  - Centre Antoine Lacassagne, Nice
  - CHU de Nîmes, Nîmes
  - CHR de la Source, Orléans
  - Hopital Saint Antoine, Paris
  - APHP - Hôpital Saint Louis, Paris
  - Hôpital de la Pitié Salpêtrière, Paris
  - APHP - Hôpital Necker, Paris
  - CH de Perpigan, Perpignan
  - CHU du Haut Leveque, Pessac
  - Clinique Francheville, Périgueux
  - CH Périgueux, Périgueux
  - Chu Lyon Sud, Pierre-Bénite
  - CHU de Poitiers, Poitiers
  - CH René Dubos, Pontoise
  - CH de Cornouaille, Quimper
  - CHU Robert Debre, Reims
  - CHU de Rennes, Rennes
  - CH de Roubaix, Roubaix
  - Centre Henri Becquerel, Rouen
  - CH de Saint Brieuc, Saint-Brieuc
  - Centre René Huguenin - Institut Curie, Saint-Cloud
  - Groupe Hospitalier Sud Réunion, Saint-Pierre
  - CH Saint Quentin, Saint-Quentin
  - CHU de Saint Malo, St-Malo
  - Strasbourg Oncologie Libérale, Strasbourg
  - CHU de Strasbourg, Strasbourg
  - CHI Toulon La Seyne-sur-mer, Toulon
  - CHU Purpan - Toulouse, Toulouse
  - CHRU Bretonneau, Tours
  - Hôpital de Valence, Valence
  - CHU de Brabois, Vandœuvre-lès-Nancy
  - CH de Bretagne Atlantique, Vannes

IPD SHARING:
Plan to Share IPD: No